CLINICAL TRIAL: NCT06757647
Title: Prospective Phase 2 Study of the Effect of Acalabrutinib on Myocardium on Ibrutinib Exposed Patients With CLL
Brief Title: Acalabrutinib for the Treatment of Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seema Bhat (Other)
Collaborators: Acerta Pharma, LLC (Other); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Seema Bhat, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23058; NCI-2024-10481 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; Specimen Handling; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (acalabrutinib) (Experimental): Patients receive acalabrutinib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CMR, CT, bone marrow aspiration/biopsy, and collection of blood samples throughout the trial.
  Interventions: Drug: Acalabrutinib; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging of the Heart

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP 196; ACP-196; ACP196; Bruton Tyrosine Kinase Inhibitor ACP-196
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging of the Heart — Undergo CMR
  Other Names: Cardiac MRI; Heart MRI

SUMMARY:
This phase II trial tests how well acalabrutinib works in treating patients with chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) and evaluates how treatment with acalabrutinib affects heart function. Acalabrutinib is in a class of medications called kinase inhibitors. It blocks a protein called BTK, which is present on B-cell (a type of white blood cells) cancers at abnormal levels. This may help keep cancer cells from growing and spreading. CLL/SLL patients treated with a different BTK inhibitor called ibrutinib often experience cardiac side effects, leading to discontinuation of life-saving therapy. Treatment with acalabrutinib after discontinuing, or even before starting, treatment with ibrutinib may reverse or prevent cardiac side effects and be an effective treatment option for patients with CLL/SLL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine cardiac magnetic resonance imaging (MRI) changes over time in patients with CLL who are intolerant to ibrutinib and switch to acalabrutinib therapy.

SECONDARY OBJECTIVES:

I. To determine the rate of recurrence of >= grade 2 adverse events (AEs) causing ibrutinib intolerance at 1 year when patients with CLL/SLL are treated with acalabrutinib.

II. To determine the response rates which include (complete response [CR], partial response [PR], PR with lymphocytosis).

III. To determine C481S/PLCG2 mutation free (defined 0 mutation bearing alleles) and clinical progression free survival at 3 years.

IV. To assess atrial fibrillation (AF) rates at 12 months post acalabrutinib transition.

EXPLORATORY OBJECTIVES:

I. To determine cardiac injury (i.e., troponin-TnT and N-terminal pro B-type natriuretic peptide [NT-proBNP]), C-reactive protein (CRP), and pro-inflammatory (ex. interleukin [IL]-6, IL-17, and tumor necrosis factor [TNF]-α, etc.) biomarkers.

II. To assess fibrosis, serum procollagen type I carboxy-terminal propeptide (PICP), galectin-3, transforming growth factor (TGF)-β1, and matrix metalloproteinases (MMPs)-2, and -7 will be collected and measured at each timepoint.

III. To determine cardiac magnetic resonance imaging (CMR) imaging changes that may be induced by acalabrutinib over time in BTK naive patients.

OUTLINE:

Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CMR, computed tomography (CT), bone marrow aspiration/biopsy, and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >= 18 years of age
* Diagnosis of CLL/SLL meeting criteria as defined by International Workshop on Chronic Lymphocytic Leukemia (iWCLL) 2018 criteria
* CLL patients cardiac intolerant to current treatment with ibrutinib as defined by AF or other cardiac arrhythmias. Other ibrutinib-related intolerances will be excluded
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Absolute neutrophil count (ANC) >= 1000/mm^3 (Independent of growth factor support at screening unless due to marrow involvement by CLL/SLL and/or disease-related immune thrombocytopenia. If cytopenias are due to disease in the bone marrow any degree of cytopenias is allowed. Patients with active uncontrolled autoimmune cytopenias are excluded)
* Platelets >= 30,000/mm^3 (Independent of growth factor support at screening unless due to marrow involvement by CLL/SLL and/or disease-related immune thrombocytopenia. If cytopenias are due to disease in the bone marrow any degree of cytopenias is allowed. Patients with active uncontrolled autoimmune cytopenias are excluded)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (excepting Gilbert's syndrome) (at screening)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN (at screening)
* Creatinine clearance >= 30 mL/min/1.73m^2 (at screening)

  * Using 24-hour creatinine clearance or modified Cockcroft-Gault equation
* Woman of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and for 2 days after the last dose of acalabrutinib
* Willing and able to participate in all required evaluations and procedures in this study protocol
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information

Exclusion Criteria:

* Prior exposure to acalabrutinib for primary cohort and prior exposure to BTK inhibitor for pilot cohort
* Presence of C481S mutation or PCLG2 mutation
* Disease progression on ibrutinib
* History of prior malignancy that could affect compliance with the protocol or interpretation of results, except for the following:

  * Curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or carcinoma in situ of the prostate at any time prior to study
  * Other cancers not specified above that have been curatively treated by surgery and/or radiation therapy from which subject is disease-free for >= 3 years without further treatment
* Clinically significant cardiovascular disease such as prior myocarditis, congestive heart failure, prior documented myocardial infarction (i.e., not self-reported), known infiltrative cardiomyopathy (ex. cardiac sarcoidosis, cardiac amyloidosis, etc.) or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Note: Subjects with controlled, asymptomatic atrial fibrillation can enroll on study
* Prior allogeneic stem cell transplantation
* Prior cardiac transplantation
* Systemic or non-cancer targeted anti-inflammatory medications (i.e., steroids)
* Contradictions to MRI: non-compatible metal implant, weight > 300 pounds (lbs.) (MRI scanner limit), severe claustrophobia, advanced or end-stage renal disease (ESRD) (contraindication to gadolinium), pregnancy, cognitive disabilities that may impair ability to comply with instructions or provide informed consent
* Has difficulty with or is unable to swallow oral medication or has significant. gastrointestinal disease that would limit absorption of oral medication
* Known history of infection with HIV or any active significant infection (e.g., bacterial, viral, or fungal) including subjects with positive cytomegalovirus [CMV] deoxyribonucleic acid [DNA] polymerase chain reaction [PCR])
* Known history of hypersensitivity or anaphylaxis to study drug(s) including active product or excipient components
* Active bleeding or history of bleeding diathesis (e.g., hemophilia or von Willebrand disease)
* Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura)
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks of the first dose of study drug is prohibited
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists
* Prothrombin time (PT)/international normalized ratio (INR) or activated partial thromboplastin time (aPTT) (in the absence of lupus anticoagulant) > 2 x ULN
* Requires treatment with proton pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Note: Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study
* History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug
* Major surgical procedure within 28 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug
* Received a live virus vaccination within 28 days of first dose of study drug
* History of or ongoing confirmed progressive multifocal leukoencephalopathy (PML)
* Received any investigational drug within 30 days or 5 half-lives (whichever is shorter) before first dose of study drug
* Hepatitis B or C serologic status:

  * Subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative polymerase chain reaction (PCR) and must be willing to undergo DNA PCR testing during the study to be eligible. Those who are HBsAg positive or hepatitis B PCR positive will be excluded
  * Subjects who are hepatitis C antibody positive will need to have a negative PCR result to be eligible. Those who are hepatitis C PCR positive will be excluded
* Breastfeeding or pregnant
* Concurrent participation in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac magnetic resonance imaging changes | Baseline to 3-month post acalabrutinib initiation
  The cardiac MRI changes that will be assessed include Extracellular volume (ECV), Native T1, and T2, where changes in ECV from baseline to 3-month post acalabrutinib initiation would be the primary endpoint

SECONDARY OUTCOMES:
Overall response rate (ORR) | At the end of cycle 24 (1 cycle = 28 days)
  ORR will be defined as the number of patients with a response (complete response [CR], partial response [PR], PR with lymphocytosis) divided by the number of eligible patients who start study treatment. Response rates including CR and ORR will be estimated at the end of treatment and at various time points with exact 95% confidence intervals. The change in response over time will be presented in a descriptive manner as well as graphically through use of a Sankey plot.
Clinical progression free survival (PFS) | From start of study treatment until first progression or death, assessed at 3 years
  PFS will be described using the method of Kaplan-Meier and estimates at 3 years will be provided with 95% confidence intervals.
C481S/PLCG2 mutation free survival | At 3 years
  Mutation free survival will be described using the method of Kaplan-Meier and estimates at 3 years will be provided with 95% confidence intervals.
Incidence of recurrence of grade 2 or greater adverse events (AEs) that previously led to ibrutinib intolerance | During the first 12 cycles of single agent acalabrutinib (1 cycle = 28 days)
  The recurrence rate will be calculated as the number of patients who have recurrence (grade 2 or higher) of the AE that previously led to ibrutinib intolerance during the first 12 cycles of single agent acalabrutinib therapy divided by the number of eligible patients who start acalabrutinib therapy. The rate of recurrence of grade 2 or greater AEs will be analyzed using an exact binomial test for a single proportion and will be estimated with exact 95% confidence intervals.
Atrial fibrillation (AF) rates | At 12 months post acalabrutinib transition
  AF rates will be calculated as the number of patients having AF (any grade) during the first 12 cycles of single agent acalabrutinib divided by the number of eligible patients who start acalabrutinib therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Seema A Bhat, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu